CLINICAL TRIAL: NCT01822886
Title: Phase IIa Study on the Role of Gemcitabine Plus Romidepsin (GEMRO Regimen) in the Treatment of Relapsed/Refractory Peripheral T-cell Lymphoma Patients.
Brief Title: Phase II Study of Gemcitabine+Romidepsin in the Relapsed/Refractory Peripheral T-cell Lymphoma Patients
Acronym: FIL_GEMRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_GEMRO
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2018-08

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: T-cell lymphoma; Romidepsin
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — romidepsin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin, Gemcitabine (Experimental): Romidepsin 12 mg/m2 day 1,8, 15 + Gemcitabine 800 mg/m2 day 1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 day 1, 15 to PD (progression disease)
  Interventions: Drug: Romidepsin + Gemcitabine

INTERVENTIONS:
Drug: Romidepsin + Gemcitabine — Romidepsin 12 mg/m2 day 1,8, 15 + Gemcitabine 800 mg/m2 day 1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 day 1, 15 to PD

SUMMARY:
Pilot clinical trial - Phase 2a, multicenter, single arm, open label trial - to evaluate efficacy and safety of concomitant combination treatment with Gemcitabine and Romidepsin (GEMRO) regimen as salvage treatment in relapsed/refractory PTCL (peripheral T-cell lymphoma) in a selected population of patients.

DETAILED DESCRIPTION:
Objectives will be focused on preliminary dose-response, type of patients, frequency of dosing, and safety and tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of PTCL according to the WHO (World Health Organization) classification
* Age ≥ 18 years
* Relapsed (≥1) or refractory to conventional chemotherapy/radiotherapy
* Stage I-IV according to the Ann Arbor staging System
* ECOG (Eastern Cooperative Oncology Group) Performance status ≤2
* Normal renal and hepatic functions
* Laboratory test results as follows:

  * Serum creatinine ≥ 2.0 mg/dL
  * Total bilirubin ≥ 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) £2 x ULN or £5 x ULN if hepatic metastases are present
  * Negative HIV HCV and HBV status
* Adequate bone marrow reserve: Platelet count>100X109 cells/L or platelet count <75X109 cells/L if bone marrow disease involvement, absolute neutrophile count (ANC)> 1,5 X109, hemoglobin>8 g/dl.
* Able to adhere to the study visit schedule and other protocol requirements
* Cardiac ejection fraction (MUGA scan or echocardiography) > 45%
* Life expectancy > 6 months
* Females of childbearing potential (FCBP) must have a negative serum or urine β-hCG pregnancy test result within 7 days prior to the first dose of study drug. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Both females of childbearing potential and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days after the last dose of study drug.
* Measurable disease of at least 2 cm as detected by CT scan, assessed by site radiologist
* Patients or they legally authorized representative must provide written informed consent

Exclusion Criteria:

* Any serious active disease or co-morbid medical condition (according to investigator's decision)
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Patients with congenital long QT syndrome, history of significant cardiovascular disease and/or taking drugs leading to significant QT prolongation
* Corrected QT interval > 480 msec (using the Fridericia formula)
* Low K+ (<3.8 mmol/L) and low Mg+ (<0.85 mmol/L) levels, except if corrected before beginning the chemotherapy
* Pregnant or lactating females or men or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study
* Previous exposure to romidepsin or gemcitabine
* CNS disease (meningeal and/or brain involvement by lymphoma) or testicular involvement
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
* Active opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, Principal Investigator — Istituto Ematologia e Oncologia Medica "SERAGNOLI" Università di Bologna
Locations (4):
- Italy (4):
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Istituto di Ematologia ed Oncologia Medica A. Seragnoli Policlinico S. Orsola, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A.O. Universitaria Citta' Della Salute E Della Scienza Di Torino, Torino

REFERENCES:
- [Derived] Pellegrini C, Dodero A, Chiappella A, Monaco F, Degl'Innocenti D, Salvi F, Vitolo U, Argnani L, Corradini P, Zinzani PL; Italian Lymphoma Foundation (Fondazione Italiana Linfomi Onlus, FIL). A phase II study on the role of gemcitabine plus romidepsin (GEMRO regimen) in the treatment of relapsed/refractory peripheral T-cell lymphoma patients. J Hematol Oncol. 2016 Apr 12;9:38. doi: 10.1186/s13045-016-0266-1. PMID 27071522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: date of first enrollment: 08 Jan 2013 date of last completed:15 Jul 2018
Groups:
- Romidepsin, Gemcitabine: Romidepsin 12 mg/m2 d.1,8, 15 + Gemcitabine 800 mg/m2 d.1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 d. 1, 15 to PD (progressioni disease)
  Romidepsin, Gemcitabine: Romidepsin 12 mg/m2 d.1,8, 15 for 6 cycles + Gemcitabine 800 mg/m2 d.1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 d. 1, 15 to PD.
Period: Overall Study
Arm/Group | Romidepsin, Gemcitabine
Started | 20
Completed | 5
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Romidepsin, Gemcitabine: Romidepsin 12 mg/m2 d.1,8, 15 + Gemcitabine 800 mg/m2 d.1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 d. 1, 15 to PD
  Romidepsin, Gemcitabine: Romidepsin 12 mg/m2 d.1,8, 15 for 6 cycles + Gemcitabine 800 mg/m2 d.1, 15 for 6 cycles by 28 days followed by Romidepsin 14 mg/m2 d. 1, 15 to PD.
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Italy | 20

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: Complete Remission is disappearance of all target lesions per the Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007)"
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
Participants | 3

2. Secondary Outcome: Percentage of Participants With Progression-Free Survival
Description: The time from start of study treatment to first documentation of objective tumor progression or to death due to any cause, whichever comes first. PFS (progression-free survival) data will be censored on the day following the date of the last radiological assessment of measured lesions documenting absence of progressive disease for patients who do not have objective tumor progression and are still on study at the time of an analysis, are given antitumor treatment other than the study treatment or stem cell transplant, or are removed from study prior to documentation of objective tumor progression. Patients lacking an evaluation of tumor response after their first dose will have their event time censored at 1 day. Percentage of participants is an estimate based on Kaplan-Meier method.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of partecipants
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
percentage of partecipants | 11.2 [3 to 25]

3. Secondary Outcome: Overall Survival is Measured From the Date of Study Entry to the Date of Patient's Death
Description: OS (overall survival) is measured from the date of study entry to the date of patient's death. If the patient is alive or his vital status is unknown, the date of death will be censored at the date that the patient is last known to be alive.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of partecipants
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
percentage of partecipants | 50 [28 to 72]

4. Secondary Outcome: Safety - Frequency of Toxicities Grade 3 and 4
Description: Frequency of toxicities was reported by type and grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0).
Time Frame: 24 months
Measure: Number; unit: events
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
events | 29

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR the proportion of patients who achieve CR (complete response), CRu (complete remission unconfirmed) or PR (partial response) relative to the per-protocol population. Disease response and progression will be evaluated according to the "Revised Response Criteria" for malignant lymphoma (Cheson et al. 2007).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Romidepsin, Gemcitabine
Number analyzed (Participants) | 20
Participants | 6

ADVERSE EVENTS:
Arm/Group | Romidepsin, Gemcitabine
All-Cause Mortality (participants affected / at risk) | 10/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Romidepsin, Gemcitabine (N=20)
Fever with shiver, Hypotension, Desaturation (General disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever, loss of consciousness and urinary infection (Renal and urinary disorders) | 1 (1)
Fever and pulmonary insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Ischaemic encephalopaty (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Romidepsin, Gemcitabine (N=20)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Nausea and vomiting (Gastrointestinal disorders) | 10 (10)
Pyrexia (General disorders) | 6 (6)
Transaminases increase (Hepatobiliary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No